CLINICAL TRIAL: NCT04220359
Title: Early Identification of Hospitalized Patients at High-risk for Clinical Deterioration During the First 72-hours in an Internal Medicine Department. A Prospective, Continuous, Physiologic Big-data-analysis Study
Brief Title: Early Identification of Clinical Deterioration Using a Wearable Monitoring Device
Status: Completed | Type: Observational
Sponsor: Biobeat Technologies Ltd. (Industry)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: Biobeat005
Record Dates: First submitted 2020-01-01; First posted 2020-01-07 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Clinical Deterioration; Hemodynamic Instability
Keywords: vital signs; clinical deterioration; early prediction; non-invasive monitoring
MeSH Terms: conditions — Clinical Deterioration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: non-invasive monitoring — Prospective monitoring with retrospective big-data analysis
  Other Names: BB-613PW

SUMMARY:
This study aims to provide myriad of physiological parameters in patients admitted in an internal medicine department, and which are defined as being in an increased risk of clinical deterioration within the first 72-hours after admission. The investigators will also conduct a retrospective comparison between physiological changes in patients who did deteriorate to those who did not. This will form the basis for the development of an algorithm for early prediction and warning of physiological and clinical deterioration during the first 72-hours of admission.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 18 years old and above admitted to the internal medicine department
* On admission, the primary investigator assess their risk to deteriorate during the first 72 hours after admission as reasonably high
* The patient is assigned to a "monitoring bed" within the department
* The patient has signed an informed consent form

Exclusion Criteria:

* Lack of informed consent
* It is known in advance that the patient cannot take part in the study for a 72-hours period (e.g. a patient that will be taken to surgery within the next 24 hours)
* Technical inability to attach the Biobeat patch (BB-613PW) to the patients chest

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients 18 years and older admitted to the internal medicine department and are at high-risk for clinical deterioration during the first 72-hours after admission. The investigators anticipate it will include patients with acute and chronic cardio-respiratory disease, systemic infections, etc.
Sampling Method: Non-Probability Sample
Enrollment: 410 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Monitoring blood pressure changes in high-risk patients | 72 hours per individual
  The investigators will record blood pressure measurements using a non-invasive wireless monitoring device working continuously for 72 hours in high-risk patients.

SECONDARY OUTCOMES:
Monitoring early heart rate changes in high-risk patients | 72 hours per individual
  The investigators will record heart rate using a non-invasive wireless monitoring device working continuously for 72 hours in high-risk patients.
Monitoring respiratory rate changes in high-risk patients | 72 hours per individual
  The investigators will record respiratory rate using a non-invasive wireless monitoring device working continuously for 72 hours in high-risk patients.
Monitoring blood oxygen saturation changes in high-risk patients | 72 hours per individual
  The investigators will record blood oxygen saturation using a non-invasive wireless monitoring device working continuously for 72 hours in high-risk patients.
Monitoring stroke volume changes in high-risk patients | 72 hours per individual
  The investigators will record stroke volume measurements using a non-invasive wireless monitoring device working continuously for 72 hours in high-risk patients.
Monitoring cardiac output changes in high-risk patients | 72 hours per individual
  The investigators will record cardiac output measurements using a non-invasive wireless monitoring device working continuously for 72 hours in high-risk patients.

CONTACTS AND LOCATIONS:
Overall Officials: Gad Segal, MD, Principal Investigator — The Sheba Medical Center, Tel Hashomer, Ramat Gan, Israel
Locations (1):
- The Sheba Medical Center, Tel Hashomer, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided
The investigators plan to publish the data in a way that will allow all readers to access the data collected and analyzed

REFERENCES:
- [Derived] Itelman E, Shlomai G, Leibowitz A, Weinstein S, Yakir M, Tamir I, Sagiv M, Muhsen A, Perelman M, Kant D, Zilber E, Segal G. Assessing the Usability of a Novel Wearable Remote Patient Monitoring Device for the Early Detection of In-Hospital Patient Deterioration: Observational Study. JMIR Form Res. 2022 Jun 9;6(6):e36066. doi: 10.2196/36066. PMID 35679119